CLINICAL TRIAL: NCT06098066
Title: Decoding the Surgical Enigma: A Groundbreaking Nationwide Study Unveils the Risks and Rewards of EC-IC Bypass, CEA, and CAS in Ischemic Cerebrovascular Disease
Brief Title: Decoding Risks and Rewards in Ischemic Stroke Surgery
Status: Completed | Type: Observational
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, XianXiu Chen, Clinical Researcher, China Medical University Hospital
Other Study IDs: NS01
Record Dates: First submitted 2023-10-09; First posted 2023-10-24 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Ischemic Stroke
Keywords: Ischemic Cerebrovascular Disease; EC-IC Bypass; Carotid Endarterectomy; Carotid Artery Stenting; Nationwide Cohort Study; Risk-Benefit Analysis
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- control
- ECIC bypass
- CEA
- CAS

SUMMARY:
In the high-stakes battle against ischemic cerebrovascular disease, where every second counts and the margin for error is slim, how do the investigators tip the scales in favor of patient survival and improved outcomes? This groundbreaking study, the first nationwide, population-based analysis with long-term follow-up in an Asian context, dives deep into this critical question. Leveraging an expansive dataset from Taiwan's National Health Insurance Research Database, the investigators scrutinize the efficacy and risks of aggressive surgical interventions-specifically, EC-IC bypass, CEA, and CAS-in a cohort of over 84,000 patients.

This paper serves as a milestone, bridging the gap between medical idealism and clinical reality. It calls for a surgical renaissance, emphasizing the need for refining techniques and enhancing patient selection protocols. If participants're looking for a comprehensive, nuanced, and, above all, actionable insight into the surgical treatment of ischemic cerebrovascular disease, this is the study that could redefine the paradigm.

ELIGIBILITY:
Inclusion Criteria:

- All participants underwent either a computed tomography (CT) scan or magnetic resonance imaging (MRI) within two days before or after hospital admission.

The date of the first ischemic stroke hospitalization served as the index event.

Among these patients, those who underwent surgical interventions post-hospitalization were categorized into three distinct groups: CEA (ICD-9-CM code 3812), CAS (ICD-9-CM code 3990), and EC-IC (ICD-9-CM code 3928), with the operation date being the index date.

Those who did not receive any surgical interventions were considered the non-intervention control group and had their first hospitalization date as the index date.

Exclusion Criteria:

- patients with a history of: any stroke subtype (ICD-9-CM codes 430-434), Moyamoya disease (ICD-9-CM code 437.5), cancer (ICD-9-CM codes 140-239), trauma (various ICD-9-CM codes), transient ischemic attack (ICD-9-CM code 435), unruptured cerebral aneurysm (ICD-9-CM code 437.3), or subarachnoid hemorrhage (ICD-9-CM code 430).

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The cohort comprises all inpatients hospitalized between January 1, 2001, and December 31, 2010, diagnosed with a first stenosis-occlusion ischemic stroke (ICD-9-CM codes 433-434). All participants underwent either a computed tomography (CT) scan or magnetic resonance imaging (MRI) within two days before or after hospital admission.
Sampling Method: Probability Sample
Enrollment: 204411 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
rehospitalization | Follow-up assessments were planned at 3 months, 6 months, 1 year, 2 years, and 3 years post-index date
  rehospitalization due to ischemic or hemorrhagic stroke

SECONDARY OUTCOMES:
Cardiac events | Follow-up assessments were planned at 3 months, 6 months, 1 year, 2 years, and 3 years post-index date
  congestive heart failure and acute myocardial infarction were also monitored throughout the study period.

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan